CLINICAL TRIAL: NCT02367690
Title: Phase 1/2, Multi-Dose, Evaluator-Blinded, Randomized, Vehicle & Standard Of Care-Controlled Dose-Escalation Study To Assess Safety, Tolerability, Pharmacokinetics Of Topical Selinexor In Patients With Diabetic Foot Ulcers
Brief Title: Study of Safety, Tolerability, and Pharmacokinetics of Topical Selinexor (KPT-330) Diabetic Foot Ulcer (DFU) Patients
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to enrollment challenges & improved SOC during run-in phase; no patients received KPT-330. Withdrawal is not a consequence of any safety concern.
Sponsor: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KCP-330-501
Record Dates: First submitted 2015-02-09; First posted 2015-02-20 (Estimated); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Diabetic Foot Ulcers
Keywords: Diabetes; Foot Ulcers; DFU; KPT-330; Selinexor; Karyopharm
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Foot Ulcer | interventions — selinexor; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1 (Experimental): Cohort 1 will be randomized to one of the following treatment groups:
  a) Standard-of-care (SOC) + Selinexor gel, 10 μM
  , b) SOC + vehicle gel c) SOC alone.
  Interventions: Drug: Selinexor; Other: Standard-of-Care; Other: Vehicle Gel
- Cohort 2 (Experimental): Cohort 2 will be randomized to one of the following treatment groups:
  1. Standard-of-care (SOC) + Selinexor gel, 30 μM
  2. SOC + vehicle gel
  3. SOC alone.
  Interventions: Drug: Selinexor; Other: Standard-of-Care; Other: Vehicle Gel
- Cohort 3 (Experimental): Cohort 3 will be randomized to one of the following treatment groups:
  1. Standard-of-care (SOC) + Selinexor gel, 70 μM
  2. SOC + vehicle gel
  3. SOC alone.
  Interventions: Drug: Selinexor; Other: Standard-of-Care; Other: Vehicle Gel

INTERVENTIONS:
Drug: Selinexor — Topical gel
  Other Names: KPT-330
Other: Standard-of-Care — Surgical debridement, sterile saline rinses, and dressing changes.
  Other Names: SOC
Other: Vehicle Gel — Topical vehicle gel with no active ingredients.

SUMMARY:
Patients with eligible diabetic foot ulcers will be screened, treated, and followed for complete ulcer closure. This is a randomized trial. All patients will receive standard-of-care treatment. Additionally, some patients will receive treatment with topical Selinexor gel and some will receive topical placebo gel.

DETAILED DESCRIPTION:
Approximately 30 patients who meet the eligibility criteria will be enrolled. Eligible patients with diabetic foot ulcers will be screened, randomized, treated, and followed for complete ulcer closure.

After screening, qualified patients will be treated for up to 12 weeks. Patients who achieve complete ulcer closure will be followed for an additional 12 weeks.

All patients will receive standard-of-care treatment. After randomization some patients will be treated with topical Selinexor gel twice weekly and some patients will be treated with a topical placebo gel twice weekly. Patients receiving Selinexor will be assigned to a sequential treatment cohort, either a 10 μM (μmol/L), 30 μM, or 70 μM dose.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a clinical diagnosis of Type I or Type II diabetes mellitus with an HbA1c ≤ 10.0 and has a BMI ≤40.
* The DFU(s) to be treated must be:

  * Anatomically discrete,
  * Non-healing, but has persisted for ≤12 months
  * Measures 1 cm2 ≤ area ≤ 5 cm2 following debridement,
  * Has a Wagner Grade 1 (i.e., not involving bone, muscle, tendons, or ligaments),
  * The Target DFU is located distal to the ankle (i.e., below the malleolus), and
  * Is able to be adequately off-loaded.
* The patient has adequate arterial blood supply in the affected limb at screening.
* Patient has the inability to perceive 10 grams pressure in the peri-ulcer area and other regions of the affected foot and toes using Semmes-Weinstein 5.07 monofilament at screening.

Exclusion Criteria:

* Patient has a foot ulcer that is clearly of non-diabetic pathophysiology.
* Patient has more than two (2) DFUs on the target lower extremity.
* DFU is clinically infected.
* Patient has active osteomyelitis of the foot or active, uncontrolled, connective tissue disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2015-05 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Presence of Local Skin Reactions (LSR) | 84 days
  Presence of local skin reactions (erythema, edema, pain, tenderness, induration, swelling, wound drainage, purulence, odor, cellulitis, callus, and maceration) within 4 cm of the diabetic foot ulcer wound edge.

SECONDARY OUTCOMES:
Ulcer Closure | 84 days
  Proportion of patients in each treatment group with complete ulcer closure of the target diabetic foot ulcer.

CONTACTS AND LOCATIONS:
Locations (1):
- South Pacific Clinical Trials, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: Yes